CLINICAL TRIAL: NCT01415921
Title: Augmentation of Parasympathetic Signaling With Pyridostigmine in Heart Failure
Brief Title: Safety Study of Pyridostigmine in Heart Failure
Acronym: APP-HF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Nathan Kline Institute for Psychiatric Research (Other); Oklahoma State University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-02167; 10-02167 (Other: NYU IRB); 1R01HL103988 (NIH)
Record Dates: First submitted 2011-08-10; First posted 2011-08-12 (Estimated); Results first posted 2016-10-25 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Heart Failure
Keywords: heart failure; autonomic function; sympathovagal balance; cholinesterase inhibitors; pharmacology
MeSH Terms: conditions — Heart Failure | interventions — Pyridostigmine Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pyridostigmine Bromide (Experimental): Forced titration protocol 15-60 mg every 8 hours as tolerated
  Interventions: Drug: Pyridostigmine Bromide
- Placebo (Placebo Comparator): Matching placebo forced titration 15-60 mg as tolerated
  Interventions: Drug: Pyridostigmine Bromide

INTERVENTIONS:
Drug: Pyridostigmine Bromide — 15, 30, and 60 mg tabs, 1 tab every 8 hours for 10 weeks. Forced titration protocol increases dose at 2 week intervals from 15 to 30 to 60 mg as tolerated. Continue maximally tolerated dose for 4 weeks and then downtitrate at weekly intervals (60 to 30 to 15) and then discontinue.
  Other Names: Mestinon

SUMMARY:
Heart failure, a common heart disease affecting nearly 6 million Americans, is associated with high rates of hospitalization and death. Abnormalities in the autonomic nervous system are thought to play an important role in the progression of heart failure. This proposal aims to determine whether novel application of pyridostigmine, a drug currently approved by the FDA only for the treatment of neuromuscular disease, can improve autonomic nervous system function in heart failure patients.

DETAILED DESCRIPTION:
Autonomic dysregulation of the cardiovascular system, characterized by heightened sympathetic activity and withdrawal of parasympathetic activity promotes progression of heart failure. Pharmacological blockade of sympathetic overactivity is associated with reduced mortality risk, but there are few data on pharmacologic augmentation of parasympathetic withdrawal. Acetylcholinesterase inhibitors augment parasympathetic neurotransmission by blocking the enzymatic breakdown of acetylcholine at cholinergic receptor sites. Pyridostigmine is a short-acting, reversible acetylcholinesterase inhibitor approved by the FDA for the treatment of myasthenia gravis. Investigators propose a Phase II prospective randomized, double-blind trial to compare 12 weeks of treatment with ascending doses of pyridostigmine (15, 30, and 60 mg every 8 hours) vs. matching placebo in 60 patients with symptomatic chronic heart failure associated with left ventricular systolic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-75 years
* Symptomatic NYHA Class II-III heart failure >6 months
* Left ventricular ejection fraction <35%
* Previous implantation of implantable cardiovertor defibrillator or pacemaker
* Guideline-recommended heart failure treatment for > 3 months
* Able and willing to provide written informed consent

Exclusion Criteria:

* Contraindications to cholinergic stimulation
* Heart failure primarily attributable to genetic, valvular, infiltrative diseases
* Persistent atrial fibrillation
* Sick sinus syndrome
* Pacemaker dependency during exercise
* Severe chronotropic incompetence with peak exercise heart rate < 100 min-1
* Severe exercise intolerance (unable to complete first stage of Bruce Protocol)
* Coronary or cerebral atherothrombotic events within the past year
* Hospitalization of emergency room visit for heart failure within last 3 months
* ICD shock in last 6 months
* Diabetes mellitus with peripheral neuropathy
* Autonomic or peripheral neuropathy of any cause
* Systolic blood pressure <90 or >160 mmHg
* Resting heart rate <60 or >100 min-1
* Serum sodium < 132 mmol/L
* Serum creatinine >2.5 mg/dl
* Liver function tests >3 times upper limit of normal
* Severe anemia (Hemoglobin <10 gm/dl)
* FEV1.0 < 60% of predicted or FEV1.0/FVC ratio <70%
* PR interval >240 msec or second or third degree heart block on electrocardiogram
* Exercise limited primarily by angina or non-cardiac co-morbid condition
* Pregnant or breast-feeding women
* Current treatment with medications known to interact with pyridostigmine
* Known intolerance of oral preparations containing bromides
* Any condition (e.g., psychiatric illness or active substance abuse) or situation that, in the investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's ability to adhere with study procedures.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart D Katz, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Langone Medical Center, New York, New York, United States

REFERENCES:
- [Background] Androne AS, Hryniewicz K, Goldsmith R, Arwady A, Katz SD. Acetylcholinesterase inhibition with pyridostigmine improves heart rate recovery after maximal exercise in patients with chronic heart failure. Heart. 2003 Aug;89(8):854-8. doi: 10.1136/heart.89.8.854. PMID 12860856
- [Derived] Goldberg R, Norcliffe-Kaufmann L, Kaufmann H, Jeschke-Lopez I, Guo Y, Zhong J, Berger KI, Goldring RM, Goldstein DS, Pope C, Maxwell L, Bharadwaj M, Reyentovich A, Katz SD. Pharmacodynamics, Safety, and Tolerability of Pyridostigmine Bromide in Heart Failure. Curr Ther Res Clin Exp. 2025 Oct 31;103:100814. doi: 10.1016/j.curtheres.2025.100814. eCollection 2025. PMID 41357360

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Admissions logs and other existing electronic hospital information systems
Period: Overall Study
Arm/Group | Pyridostigmine Bromide | Placebo
Started | 16 | 17
Completed | 13 | 14
Not Completed | 3 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pyridostigmine Bromide | Placebo | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 15 | 29
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 14 | 15 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 2 | 0 | 2
  More than one race | 8 | 9 | 17
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Baseline Heart Rate Recovery
Description: Change in peak HR at end of exercise to 1 minute post-exercise (beats per minute)
Time Frame: Baseline
Population: Heart rate recovery is also measured as beats/min (peak HR at end of exercise - HR 1 min post exercise = HRR).
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Pyridostigmine Bromide | Placebo
Number analyzed (Participants) | 13 | 14
beats per minute | 32.5 (12.8) | 30.4 (14.8)

2. Primary Outcome: Post Exercise Heart Rate Recovery
Description: Change in heart rate from peak exercise to 1 minute post-exercise (beats per minute)
Time Frame: 12 weeks
Population: Heart rate recovery is also measured as beats/min (peak HR at end of exercise - HR 1 min post exercise = HRR).
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Pyridostigmine Bromide | Placebo
Number analyzed (Participants) | 13 | 14
beats per minute | 38.5 (12.2) | 34.9 (16.1)

ADVERSE EVENTS:
Arm/Group | Pyridostigmine Bromide | Placebo
Serious Adverse Events (participants affected / at risk) | 2/16 | 3/17
Other Adverse Events (participants affected / at risk) | 11/16 | 10/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pyridostigmine Bromide (N=16) | Placebo (N=17)
Decompensated Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Elective Stent Placement (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal Paim (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Ventricular Malposition of an ICD Lead (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pyridostigmine Bromide (N=16) | Placebo (N=17)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
Blurred vision of right eye (Eye disorders) | 0 (0) | 1 (1)
Loose Stools (Gastrointestinal disorders) | 2 (2) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Black Stool (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Ankle sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pacemaker AMS (Investigations) | 1 (1) | 0 (0)
Inadequate ICD shock (Investigations) | 0 (0) | 1 (1)
Ventricular pacing (Investigations) | 0 (0) | 1 (1)
Supraventicular tachycardia reported on ICD (Investigations) | 0 (0) | 1 (1)
Total Bilirubin Increased (Investigations) | 0 (0) | 1 (1)
Elevated Alkaline Phosphatase (Investigations) | 1 (1) | 0 (0)
Elevated hepatic enzymes (Investigations) | 0 (0) | 1 (1)
Thrombocitopenia (Investigations) | 0 (0) | 1 (1)
Percent Eosinophils Increased (Investigations) | 1 (1) | 0 (0)
PMT (Pacemaker Tachycardia) (Investigations) | 1 (1) | 0 (0)
Pain in lower extremities (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendinitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Plantar Fasciitis
Gout (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) — Dizziness
Urinary Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) — Urinary Incontinence
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Sore throat
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Sweating
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Rash
Low heart rate (Vascular disorders) | 1 (1) | 1 (1) — Low heart rate
Hypertension (Vascular disorders) | 0 (0) | 2 (2) — Hypertension

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes